CLINICAL TRIAL: NCT01831921
Title: Latinos Combatiendo la Diabetes (Latinos Combating Diabetes)
Brief Title: Latinos Combating Diabetes
Acronym: La Comunidad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00022566; 1P60MD006917 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pre Diabetes; Obesity; Metabolic Syndrome
Keywords: pre diabetes; obesity; weight loss; lifestyle; prevention
MeSH Terms: conditions — Glucose Intolerance; Obesity; Metabolic Syndrome; Weight Loss | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Weight-Loss (Experimental): Participants in the Behavioral: Lifestyle Weight Loss arm will take part in a group program aimed at achieving modest weight loss (5-7%) through promoting healthy eating and increasing physical activity. The intervention sessions will take place at churches and other community locations and will be coordinated and facilitated by Latino Health Advisors (LHAs). The lifestyle intervention will be delivered in 2 phases: Phase 1 will last for 6 months and consist of weekly group meetings; Phase 2 will last for 18 months and consist of one LHA-led group session or one telephone contact from the LHA per month. Participants in this treatment arm will also receive individual visits with a registered dietitian during months 1, 3, and 6 of phase 1. All participants will be seen for assessment visits as baseline, 6, and 12 months. Some participants will also complete 18 and 24 month visits, depending on the date of randomization.
  Interventions: Behavioral: Lifestyle Weight Loss
- Enhanced Usual Care (Active Comparator): Participants in the Behavioral: Counseling arm will receive two individual sessions with a registered dietitian and monthly newsletters that focus on existing community resources.All participants will be seen for assessment visits as baseline, 6, and 12 months. Some participants will also complete 18 and 24 month visits, depending on the date of randomization.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Lifestyle Weight Loss — Changing diet, physical activity, and self-regulatory behaviors to promote weight loss.
  Arms: Lifestyle Weight-Loss
Behavioral: Counseling — Individual nutrition counseling will be delivered by a registered dietitian.
  Arms: Enhanced Usual Care

SUMMARY:
The investigators plan to test two different strategies for weight loss and diabetes prevention in the Latino community in and around Forsyth County, North Carolina. The study is designed to test the hypothesis that a lifestyle weight-loss program implemented within the Latino community will have a more beneficial and clinically meaningful impact on hemoglobin A1c (HbA1c), insulin metabolism, and markers of the metabolic syndrome when compared to an enhanced usual care condition. This lifestyle intervention will include group-based sessions promoting healthy eating, increased physical activity and weight loss. These sessions will be delivered by lay community members, known as Latino Health Advisors (LHAs). The enhanced usual care group will consist of individual counseling with are registered dietitian and uses existing community resources to assist participants in making healthier lifestyle choices.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a major health concern in the United States, accounting for 90 to 95% of the more than 25 million diagnosed cases of diabetes in 2010. Racial and ethnic minorities are disproportionately affected by the diabetes epidemic, specifically African Americans, Latinos, and Native Americans. Although the cumulative evidence suggests that lifestyle interventions to prevent diabetes can be implemented across a variety of settings with diverse personnel, numerous barriers to widespread dissemination in minority populations still exist. Latinos Combatiendo la Diabetes (La Comunidad) is a 225-participant randomized trial designed to test the hypothesis that a community-based lifestyle weight-loss intervention implemented within the accountability and structure of existing Latino communities will have a more beneficial and clinically meaningful impact on HbA1c, insulin metabolism, and markers of the metabolic syndrome when compared to an enhanced usual care condition. An economic evaluation will also be conducted to determine costs and cost-effectiveness. One trial arm will consist of a group-based intensive lifestyle intervention promoting healthy eating, increased physical activity and modest, yet achievable (5-7%) weight loss delivered in an early 6-month intensive phase followed by an 18-month maintenance phase. Latino Health Advisors (LHAs) will be utilized in the intensive intervention arm. The control arm will consist of an individual educational intervention that incorporates existing community resources that are available to assist residents in making healthier lifestyle choices.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and older who reside in or near Forsyth County, North Carolina
* Self-identified as Hispanic or Latino
* Evidence of pre-diabetes: Hemoglobin A1c of 5.7-6.5%
* Body Mass Index (BMI): 25-45 kg/m2
* Potential participants must be willing to accept randomization to either the intensive lifestyle intervention or the comparison usual care condition

Exclusion Criteria:

* Currently involved in a supervised program for weight loss
* Clinical history of diabetes or newly diagnosed diabetes at screening
* Clinical history of cardiovascular disease (CVD) occurring within the past 6 months, including myocardial infarction, angina, coronary revascularization, stroke, transient ischemic attack (TIA), carotid revascularization, peripheral arterial disease, congestive heart failure. All persons with recent CVD should be participating in cardiac rehabilitation (with appropriate supervision as indicated) to reduce their risk of recurrence; hence, randomization might raise ethical concerns.
* Uncontrolled high blood pressure (BP): BP > 160/100. Potential participants can be re-screened after control has been achieved.
* Pregnancy, breast feeding, or planning pregnancy within 2 years
* Other chronic disease likely to limit lifespan to less than 2-3 years, including any cancer requiring treatment in past 5 years except non-melanoma skin cancer
* Chronic use of medicine known to significantly affect glucose metabolism (e.g., corticosteroids, protease inhibitors)
* Conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, another household member already randomized to La Comunidad, major psychiatric or cognitive problems (schizophrenia, dementia, self-reported active illegal substance or alcohol abuse), participation in another research study that would interfere with La Comunidad.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH RDN, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Baseline and randomization visits began in January 2014 and concluded in June 2016. In a roughly 26-month period, 225 participants were randomized (150 lifestyle intervention; 75 enhanced usual care) to take part in La Comunidad.
Groups:
- Lifestyle Weight-Loss: Participants in the Behavioral: Lifestyle Weight Loss arm will take part in a group program aimed at achieving modest weight loss (5-7%) through promoting healthy eating and increasing physical activity. The intervention sessions will take place at churches and other community locations and will be coordinated and facilitated by Latino Health Advisors (LHAs). The lifestyle intervention will be delivered in 2 phases: Phase 1 will last for 6 months and consist of weekly group meetings; Phase 2 will last for 18 months and consist of one LHA-led group session or one telephone contact from the LHA per month. Participants in this treatment arm will also receive individual visits with a registered dietitian during months 1, 3, and 6 of phase 1.
  Lifestyle Weight Loss: Changing diet, physical activity, and self-regulatory behaviors to promote weight loss.
- Enhanced Usual Care: Participants in the Behavioral: Counseling arm will receive two individual sessions with a registered dietitian and monthly newsletters that focus on existing community resources.
  Counseling: Individual nutrition counseling will be delivered by a registered dietitian.
Period: Overall Study
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Started | 150 | 75
6 Months | 122 | 63
12 Months | 120 (All participants were followed for 12 months to 24 months, depending on date of randomization.) | 62
18 Months | 90 (Of 118 eligible for this visit.) | 49 (Of 59 eligible for this visit.)
Completed | 66 (Of 85 eligible for this visit.) | 36 (Of 42 eligible for this visit.)
Not Completed | 84 | 39

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Usual Care: Participants in the Behavioral: Counseling arm will receive two individual sessions with registered dietitian and monthly newsletters that focus on existing community resources.
  Counseling: Individual nutrition counseling will be delivered by a registered dietitian.
- Total: Total of all reporting groups
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care | Total
Number analyzed (Participants) | 150 | 75 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 147 | 71 | 218
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (9.0) | 41.8 (9.1) | 41.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 64 | 191
  Male | 23 | 11 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 150 | 75 | 225
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 75 | 225
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 6.0 (.30) | 5.9 (.20) | 5.9 (.3)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 81.9 (14.10) | 80.3 (13.1) | 81.4 (13.80)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118.5 (13.8) | 116.5 (14.5) | 117.8 (14.0)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 71.9 (8.5) | 69.9 (9.8) | 71.3 (9.0)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 97.7 (9.9) | 96.6 (9.6) | 97.4 (9.8)
High Density Lipoprotien (HDL) [Mean (Standard Deviation); unit: mg/dL] | 45.3 (10.5) | 46.5 (10.9) | 45.7 (10.6)
Low Density Lipoprotein (LDL) [Mean (Standard Deviation); unit: mg/dL] | 109.9 (28.50) | 106.7 (28.10) | 108.8 (28.40)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 142.1 (68.70) | 140.1 (61.60) | 141.4 (66.30)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 183.6 (33.10) | 181.3 (36.6) | 182.8 (34.30)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Mean hemoglobin A1c in both treatment groups at 6, 12, 18, and 24 months will be assessed.
Time Frame: 6, 12, 18, and 24 months
Population: Participant retention at clinic assessment visits is presented below as the number analyzed at each time-point. Follow-up on all participants was at least 12 months; for those participants randomized early in the recruitment process, 18 and 24 month data was collected.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Groups:
- Lifestyle Weight-Loss: Participants in the Behavioral: Lifestyle Weight Loss arm will take part in a group program aimed at achieving modest weight loss (5-7%) through promoting healthy eating and increasing physical activity. The intervention sessions will take place at churches and other community locations and will be coordinated and facilitated by LHAs. The lifestyle intervention will be delivered in 2 phases: Phase 1 will last for 6 months and consist of weekly group meetings; Phase 2 will last for 18 months and consist of one LHA-led group session or one telephone contact from the LHA per month. Participants in this treatment arm will also receive individual visits with a registered dietitian during months 1, 3, and 6 of phase 1.
  Lifestyle Weight Loss: Changing diet, physical activity, and self-regulatory behaviors to promote weight loss.
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
percent HbA1c
  6 Months: number analyzed (Participants) | 122 | 63
  6 Months | 5.9 (.30) | 5.8 (.30)
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 5.9 (.30) | 5.9 (.30)
  18 Months: number analyzed (Participants) | 90 | 75
  18 Months | 5.9 (.30) | 5.9 (.30)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 6.0 (.40) | 6.0 (.50)

2. Secondary Outcome: Body Weight
Description: Mean body weight in both treatment groups at 6, 12, 18, and 24 months will be assessed.
Time Frame: 6, 12, 18, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Lifestyle Weight-Loss: Participants in the Behavioral: Lifestyle Weight Loss arm will take part in a group program aimed at achieving modest weight loss (5-7%) through promoting healthy eating and increasing physical activity. The intervention sessions will take place at churches and other community locations and will be coordinated and facilitated by LHAs. The lifestyle intervention will be delivered in 2 phases: Phase 1 will last for 6 months and consist of weekly group meetings; Phase 2 will last for 18 months and consist of one LHA-led group session or one telephone contact from the LHA per month. Participants in this treatment arm will also receive individual visits with an RD during months 1, 3, and 6 of phase 1.
  Lifestyle Weight Loss: Changing diet, physical activity, and self-regulatory behaviors to promote weight loss.
- Enhanced Usual Care: Participants in the Behavioral: Counseling arm will receive two individual sessions with an RD and monthly newsletters that focus on existing community resources.
  Counseling: Individual nutrition counseling will be delivered by a registered dietitian.
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
kilograms
  6 Months: number analyzed (Participants) | 122 | 63
  6 Months | 79.2 (14.3) | 77.4 (13.1)
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 79.7 (14.1) | 79.1 (13.9)
  18 Months: number analyzed (Participants) | 90 | 49
  18 Months | 79.9 (14.5) | 78.7 (13.6)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 80.0 (13.7) | 77.3 (12.2)

3. Secondary Outcome: Systolic Blood Pressure
Description: Mean systolic blood pressure in both treatment groups at 6, 12, 18, and 24 months will be assessed.
Time Frame: 6, 12, 18, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mmHg
  6 Months: number analyzed (Participants) | 122 | 63
  6 Months | 117.0 (14.5) | 113.7 (12.9)
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 116.7 (13.2) | 114.3 (11.9)
  18 Months: number analyzed (Participants) | 90 | 49
  18 Months | 117.1 (12.6) | 115.6 (12.8)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 119.7 (16.6) | 116.8 (10.7)

4. Secondary Outcome: Diastolic Blood Pressure
Description: Mean diastolic blood pressure in both treatment groups at 6, 12, 18, and 24 months will be assessed.
Time Frame: 6, 12, 18, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mmHg
  6 Months: number analyzed (Participants) | 122 | 63
  6 Months | 69.5 (9.4) | 69.2 (9.5)
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 70.0 (9.9) | 71.2 (8.9)
  18 Months: number analyzed (Participants) | 90 | 49
  18 Months | 69.3 (9.3) | 70.4 (8.1)
  24 Months: number analyzed (Participants) | 66 | 75
  24 Months | 70.5 (9.7) | 70.7 (8.4)

5. Secondary Outcome: Fasting Glucose
Description: Mean fasting plasma glucose in both treatment groups at 6, 12, 18, and 24 months will be assessed.
Time Frame: 6, 12, 18, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mg/dL
  6 Months: number analyzed (Participants) | 122 | 63
  6 Months | 96.3 (10.3) | 96.3 (8.7)
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 98.1 (10.1) | 96.1 (11.6)
  18 Months: number analyzed (Participants) | 90 | 49
  18 Months | 98.0 (11.7) | 98.6 (14.2)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 98.2 (10.5) | 99.9 (17.9)

6. Secondary Outcome: Total Cholesterol
Description: Mean total cholesterol in both treatment groups at 12 and 24 months will be assessed.
Time Frame: 12, and 24 months
Population: Participant retention at clinic assessment visits is presented below as the number analyzed at each time-point. Follow-up on all participants was at least 12 months; for those participants randomized early in the recruitment process, 24 month data was collected.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mg/dL
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 181.1 (35.5) | 180.3 (36.9)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 184.7 (40.0) | 174.4 (40.3)

7. Secondary Outcome: High Density Lipoprotein (HDL)
Description: Mean HDL in both treatment groups at 12 and 24 months will be assessed.
Time Frame: 12, and 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mg/dL
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 47.3 (11.6) | 47.5 (11.2)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 46.8 (10.5) | 45.5 (9.8)

8. Secondary Outcome: Low Density Lipoprotein (LDL)
Description: Mean LDL in both treatment groups at 12 and 24 months will be calculated.
Time Frame: 12, and 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mg/dL
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 106.7 (27.9) | 106.5 (31.8)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 108.3 (31.4) | 101.5 (25.4)

9. Secondary Outcome: Triglycerides
Description: Mean triglycerides in both treatment groups at 12 and 24 months will be calculated.
Time Frame: 12, and 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
Number analyzed (Participants) | 150 | 75
mg/dL
  12 Months: number analyzed (Participants) | 120 | 62
  12 Months | 139.7 (76.6) | 131.3 (56.7)
  24 Months: number analyzed (Participants) | 66 | 36
  24 Months | 147.7 (74.8) | 139.3 (153.9)

10. Other Pre Specified Outcome: Fasting Insulin
Description: Mean change in fasting insulin from baseline between treatment groups at 6, 12, and 24 months will be assessed.
Time Frame: 6, 12, and 24 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Homeostasis Model of Insulin Resistance (HOMA IR)
Description: Mean change in the HOMA IR model from baseline between treatment groups at 6, 12, and 24 months will be assessed.
Time Frame: 6, 12, and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events and serious adverse events was collected every 6 months for up to 24 months.
Arm/Group | Lifestyle Weight-Loss | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 2/150 | 0/75
Serious Adverse Events (participants affected / at risk) | 4/150 | 1/75
Other Adverse Events (participants affected / at risk) | 13/150 | 10/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Weight-Loss (N=150) | Enhanced Usual Care (N=75)
death from non-study related causes (colon cancer) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Participant was diagnosed with late-stage colon cancer during study and died as a result of cancer progression. This event was reviewed by the study safety officer and deemed unrelated to participation.
death from non-study related causes (aneurysm) (Vascular disorders) | 1 (1) | 0 (0) — Participant suffered a ruptured aneurysm while driving and died. This event was reviewed by the study safety officer and deemed unrelated to participation.
Inpatient hospitalization for surgery (Surgical and medical procedures) | 2 (2) | 1 (1) — 3 participants were hospitalized overnight for medical procedures unrelated to study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle Weight-Loss (N=150) | Enhanced Usual Care (N=75)
Joint/Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 (150) | 10 (75) — Pain, injury, or discomfort in knee, shoulder, or other joints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT01831921/Prot_SAP_000.pdf